CLINICAL TRIAL: NCT07208760
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Effect of L9LS on R21/Matrix-M™ Vaccine Immunogenicity
Brief Title: L9LS-R21 Interaction
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institutes of Health (NIH) (NIH); Malaria Research and Training Center (MRTC) (Unknown); Faculté de Médecine Pharmacie d'Odontostomatologie (FMOS) (Unknown); University of Sciences, Techniques, and Technologies of Bamako (USTTB) (Unknown); University of Washington (Other); Indiana University School of Medicine, Indiana University (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: 2025/183/CE/USTTB
Record Dates: First submitted 2025-09-17; First posted 2025-10-06 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- L9LS in Healthy Malian Adult with R21/Matrix-M™ starting 7 days after (Experimental): L9LS with R21/Matrix-M™ series starting 7 days after.
  Interventions: Drug: Single dose of 1800 mg L9LS SC (12mL)
- Placebo in Healthy Malian Adult with R21/Matrix-M™ starting 7 days after (Placebo Comparator): Placebo with R21/Matrix-M™ series starting 7 days after.
  Interventions: Other: Placebo 12 mL SC
- L9LS in Healthy Malian Infant with R21/Matrix-M™ starting 7 days after (Experimental): L9LS with R21/Matrix-M™ series starting 7 days after.
  Interventions: Drug: Single dose of 225 mg L9LS SC (1.5mL)
- Placebo in Healthy Malian Infant with R21/Matrix-M™ starting 7 days after (Placebo Comparator): Placebo with R21/Matrix-M™ series starting 7 days after.
  Interventions: Other: Placebo 1.5 mL SC
- L9LS in Healthy Malian Infant with R21/Matrix-M™ starting 56 days after (Experimental): L9LS with R21/Matrix-M™ series starting 56 days after.
  Interventions: Drug: Single dose of 225 mg L9LS SC (1.5mL)
- Placebo in Healthy Malian Infant with R21/Matrix-M™ starting 56 days after (Placebo Comparator): Placebo with R21/Matrix-M™ series starting 56 days after.
  Interventions: Other: Placebo 1.5 mL SC
- L9LS in Healthy Malian Infant with R21/Matrix-M™ starting 112 days after (Experimental): L9LS with R21/Matrix-M™ series starting 112 days after.
  Interventions: Drug: Single dose of 225 mg L9LS SC (1.5mL)
- Placebo in Healthy Malian Infant with R21/Matrix-M™ starting 112 days after (Placebo Comparator): Placebo with R21/Matrix-M™ series starting 112 days after.
  Interventions: Other: Placebo 1.5 mL SC

INTERVENTIONS:
Drug: Single dose of 1800 mg L9LS SC (12mL) — A human monoclonal antibody to protect against Plasmodium falciparum.
  Arms: L9LS in Healthy Malian Adult with R21/Matrix-M™ starting 7 days after
Other: Placebo 12 mL SC — Normal saline.
  Arms: Placebo in Healthy Malian Adult with R21/Matrix-M™ starting 7 days after
Drug: Single dose of 225 mg L9LS SC (1.5mL) — A human monoclonal antibody to protect against Plasmodium falciparum.
  Arms: L9LS in Healthy Malian Infant with R21/Matrix-M™ starting 112 days after; L9LS in Healthy Malian Infant with R21/Matrix-M™ starting 56 days after; L9LS in Healthy Malian Infant with R21/Matrix-M™ starting 7 days after
Other: Placebo 1.5 mL SC — Normal saline.
  Arms: Placebo in Healthy Malian Infant with R21/Matrix-M™ starting 112 days after; Placebo in Healthy Malian Infant with R21/Matrix-M™ starting 56 days after; Placebo in Healthy Malian Infant with R21/Matrix-M™ starting 7 days after

SUMMARY:
This is a randomized, double-blind, placebo-controlled trial in 2 parts evaluating the effect of 1-time administration of the monoclonal antibody (MAb) L9LS to healthy Malian participants on the immunogenicity of subsequent administration of the R21/Matrix-M™ vaccine. L9LS will be administered subcutaneously (SC) for adults and infants. The study will assess how the timing of L9LS administration impacts immunogenicity following subsequent intramuscular (IM) R21/Matrix-M™ vaccination. Twenty-four adult participants and 333 infant participants will be enrolled.

DETAILED DESCRIPTION:
In Part 1, 24 adult participants will be randomized 1:1 to receive 1800 mg of L9LS or normal saline placebo at enrollment, followed by the R21/Matrix-M™ 3-dose initial vaccine series starting on day 7. Adult participants will be followed at study visits 7 days after L9LS administration and 7 days after each R21/Matrix-M™ vaccination. If no significant safety concerns arise through 7 days after administration of the first R21/Matrix-M™ vaccine (day 14) per an interim safety review, the study will proceed to Part 2. There will also be study visits 28 and 84 days following the last R21/Matrix-M™ vaccine to assess immune responses.

In Part 2, 333 infant participants will be randomized into 1 of 3 cohorts, each with an L9LS arm and a placebo arm (2:1). The individual cohorts will differ in the timing of the R21/Matrix-M™ 3-dose initial vaccine series (7 days, 2 months, and 4 months between L9LS and first R21/Matrix-M™ respectively). Infant participants will be followed at study visits 7 days after L9LS administration and 7 days after each R21/Matrix-M™ vaccination, after which they will continue to be followed every 28 days through the fourth (booster) dose of the R21/Matrix-M™ vaccine. There will also be study visits 28 and 84 days following the last R21/Matrix-M™ vaccine to assess immune responses. Primary study assessments include medical history, physical examination, and blood collection to assess antibody responses to the R21/Matrix-M™ vaccine, L9LS pharmacokinetics (PK), anti-drug antibody (ADA) assessments, identification of Plasmodium falciparum (Pf) infection by microscopic examination of thick blood smears and reverse transcription polymerase chain reaction (RT-PCR), and other research laboratory evaluations.

ELIGIBILITY:
Inclusion Criteria:

Part 1: Healthy Adults

Individuals must meet all of the following criteria to be eligible for study participation:

1. Male aged ≥18 and ≤50 years weighing ≥50.0 and ≤100.0 kg or female aged ≥18 and ≤50 years weighing ≥45.0 and ≤90.0 kg.
2. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
3. In good general health and without clinically significant medical history.
4. Able to provide informed consent.
5. Willing to have blood samples and data stored for future research.
6. Resides in or near Sotuba, Mali, and available for the duration of the study.
7. Females of childbearing potential must be willing to use reliable contraception from 21 days prior to study day 0 through the final study visit as described below.

   1. Reliable methods of birth control include 1 of the following: confirmed pharmacologic contraceptives via parenteral delivery or intrauterine or implantable device.
   2. Nonchildbearing women will be required to report date of last menstrual period, history of surgical sterility (i.e., tubal ligation, hysterectomy) or premature ovarian insufficiency, and will have serum pregnancy test performed per protocol.

Part 2: Healthy Infants

Individuals must meet all of the following criteria to be eligible for study participation:

1. Aged ≥5 and ≤12 months at enrollment.
2. Born at ≥37 weeks gestation (at term).
3. Parent and/or guardian able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
4. In good general health and without clinically significant medical history.
5. Parent and/or guardian able to provide informed consent.
6. Willing to have blood samples and data stored for future research.
7. Resides in or near Sotuba, Mali, and available for the duration of the study.

Exclusion Criteria:

Part 1: Healthy Adults

Individuals meeting any of the following criteria will be excluded from study participation:

1. Pregnancy, as determined by a positive urine or serum beta-human choriogonadotropin test (if female).
2. Currently breastfeeding.
3. Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the prospective participant to understand and comply with the study protocol.
4. Study comprehension examination score of <80% correct or per investigator discretion.
5. Hemoglobin, WBC, absolute neutrophil, or platelet count outside the local laboratory-defined limits of normal. Individuals may be included at the investigator's discretion for "not clinically significant" values.
6. ALT or creatinine (Cr) level above the local laboratory-defined upper limit of normal. Individuals may be included at the investigator's discretion for "not clinically significant" values.
7. Infection with HIV virus.
8. Known or documented sickle cell disease by history. (Note: Known sickle cell trait is NOT exclusionary.)
9. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, endocrine, rheumatologic, autoimmune, hematological, oncologic, or renal disease by history, physical examination, and/or laboratory studies.
10. Receipt of any investigational product within the past 30 days.
11. Participation or planned participation in an interventional trial with an investigational product until the last required protocol visit. (Note: Past, current, or planned participation in observational studies is NOT exclusionary; participation in the placebo arm of the Mali adult CIS43LS MAb trial [ClinicalTrials.gov Identifier: NCT04329104] or L9LS MAb trials [NCT05816330] is NOT exclusionary.)
12. Medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
13. History of a severe allergic reaction or anaphylaxis, including history of generalized urticaria and angioedema from prior allergic reactions.
14. Hypersensitivity to the active substances or to any of the excipients included in the vaccines.
15. Hypersensitivity to hepatitis B vaccines.
16. Severe asthma (defined as asthma that is unstable or required emergent care, urgent care, hospitalization, or intubation during the past 2 years, or that has required the use of oral or parenteral corticosteroids at any time during the past 2 years).
17. Pre-existing autoimmune or antibody-mediated diseases including but not limited to: systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjögren's syndrome, or autoimmune thrombocytopenia.
18. Salivary gland disorder diagnosed by a doctor (e.g., parotitis, sialadenitis, sialolithiasis, salivary gland tumors).
19. Known immunodeficiency syndrome.
20. Known asplenia or functional asplenia.
21. Use of chronic (≥14 days) oral or IV corticosteroids (excluding topical or nasal) at immunosuppressive doses (i.e., prednisone >10 mg/day) or immunosuppressive drugs within 30 days of day 0.
22. Receipt of a live vaccine within the past 4 weeks or a killed vaccine within the past 2 weeks prior to study agent administration.
23. Receipt of immunoglobulins and/or blood products within the past 6 months.
24. Previous receipt of an investigational malaria vaccine or MAb in the last 5 years.
25. Other condition(s) that, in the opinion of the investigator, would jeopardize the safety or rights of an individual participating in the trial, interfere with the evaluation of the study objectives, or render the participant unable to comply with the protocol.

Part 2: Healthy Infants

Individuals meeting any of the following criteria will be excluded from study participation:

1. Body weight <5.5 kg.
2. Behavioral, cognitive, or psychiatric disease in the parent and/or guardian that in the opinion of the investigator affects the ability of the parent and/or guardian to understand and comply with the study protocol.
3. Any fever (≥ 37.5°C, regardless of route) or acute illness within 7 days prior to randomization.
4. Clinically significant congenital anomaly or documented or suspected serious medical illness (e.g., history of epilepsy), serious congenital anomaly, or immediate life-threatening condition in the infant that may interfere with the ability to complete study requirements, as judged by the examining clinician.
5. Prior history of a suspected or actual acute medically life-threatening event.
6. Receipt of any blood products, monoclonal or polyclonal antibody/immunoglobulin (e.g., hepatitis B immune globulin, IV immunoglobulin), or anticipated use during the study.
7. Any suspected or actual life-threatening acute or chronic illnesses known in the mother during her pregnancy.
8. Parent or guardian study comprehension examination score of <80% correct or per investigator discretion.
9. Hemoglobin, WBC, absolute neutrophil, or platelet count outside the local laboratory-defined limits of normal. Individuals may be included at the investigator's discretion for "not clinically significant" values.
10. ALT or Cr level above the local laboratory-defined upper limit of normal. Individuals may be included at the investigator's discretion for "not clinically significant" values.
11. Mother and/or infant infected with HIV.
12. Sickle cell disease by testing. (Note: Known sickle cell trait is NOT exclusionary.)
13. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, endocrine, rheumatologic, autoimmune, hematological, oncologic, or renal disease by history, physical examination, and/or laboratory studies.
14. Receipt of any investigational product within the past 30 days.
15. Participation or planned participation in an interventional trial with an investigational product until the last required protocol visit. (Note: Past, current, or planned participation in observational studies is NOT exclusionary.)
16. History of a severe allergic reaction or anaphylaxis, including history of generalized urticaria and angioedema from prior allergic reactions.
17. Hypersensitivity to the active substances or to any of the excipients included in the vaccines.
18. Hypersensitivity to hepatitis B vaccines.
19. Salivary gland disorder diagnosed by a doctor (e.g., parotitis, sialadenitis, sialolithiasis, salivary gland tumors).
20. Pre-existing autoimmune or antibody-mediated diseases including but not limited to systemic lupus erythematosus or autoimmune thrombocytopenia.
21. Known immunodeficiency syndrome.
22. Known asplenia or functional asplenia.
23. Use of chronic (≥14 days) oral or IV corticosteroids (excluding topical or nasal) at immunosuppressive doses (i.e., prednisone >10 mg/day) or immunosuppressive drugs within 30 days of day 0.
24. Previous receipt of the R21/Matrix-MTM or RTS,S/AS01 vaccine.
25. Receipt of a live or killed vaccine within the past 1 week prior to study agent administration.
26. Previous receipt of an investigational malaria vaccine or MAb.
27. Previous receipt of L9LS MAb by the mother.
28. Clinical signs of malnutrition.
29. Other condition(s) that, in the opinion of the investigator, might jeopardize the safety or rights of an individual participating in the trial, interfere with the evaluation of the study objectives, or render the participant unable to comply with the protocol.

Ages: 5 Months to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 357 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Part 1: Incidence and severity of hypersensitivity reactions | Occurring within 7 days after the administration of the first dose of the R21/Matrix-M™ vaccine.
Part 2: Total IgG anti-NANP antibody titers | 28 days after the third R21/Matrix-M™ vaccination
  Measured by ECLIA, using the Meso Scale Discovery (MSD) LLC-based automation platform

SECONDARY OUTCOMES:
Part 1a: Incidence and severity of local and systemic AEs | Occurring within 7 days after the administration of L9LS and within 7 days after administration of each dose of R21/Matrix-M™.
Part 1b: Incidence and severity of laboratory abnormalities | Occurring within 7 days after the administration of study agent.
Part 2a: Incidence and severity of local and systemic AEs | Occurring within 7 days after the administration of L9LS and within 7 days after administration of each dose of R21/Matrix-M™.
Part 2b: Incidence and severity of laboratory abnormalities | Occurring within 7 days after the administration of study agent.
Part 2c: Incidence and severity of hypersensitivity reactions | Occurring within 7 days after the administration of each dose of R21/Matrix-M™ vaccine.
Part 2d: Total IgG anti-NANP antibody titers | 84 days after the third R21/Matrix-M™ vaccination.
  Measured by ECLIA, using the Meso Scale Discovery (MSD) LLC-based automation platform
Part 2e: Detection of Anti-Drug Antibodies (ADAs) to L9LS | Through study completion, an average of 2 years.
  Measured by 3-tier MSD assay
Part 2f: Serum concentrations of L9LS | Up to 18 months.
  Measured with an L9LS anti-idiotype antibody and a MSD LLC-based automation platform

CONTACTS AND LOCATIONS:
Overall Officials: Bickey H Chang, MD, MHA, Principal Investigator — LIG/NIAID/NIH; Kassoum Kayentao, MD, MPH, PhD, Principal Investigator — MRTC/FMOS/USTTB
Locations (1):
- Sotuba Malaria Research and Training Center (MRTC), Sotouba, Mali

IPD SHARING:
Plan to Share IPD: Undecided